CLINICAL TRIAL: NCT03578523
Title: Using MRI ASL Techniques for Quantitative Measurement of Renal Haemodynamics and Structural Parameters in Acute Kidney Injury and Chronic Kidney Disease.
Brief Title: Renal MR Feasibility in Renal Disease
Acronym: REMIND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 15040
Record Dates: First submitted 2016-07-12; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Renal Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease: CKD stage 3-4 eGFR 59-20mls/min/1.73 '3 Tesla multiparametric MR: Renal MRI Scan to assess blood flow, perfusion, oxygenation and microstructure (MR T1 relaxation time and diffusion).
  Each patient will have 3 renal MRI scans. renal histopathology scoring: Blinded fibrosis scoring of renal histopathology (If biopsy performed for clinical indication) Iohexol clearance test: Blood and urine sampling around scan sessions; this will include routine patient care biochemistry and haematology panel.
  urine protein and albumin measurements, stored plasma/serum/urine for subsequent analysis.
  Iohexol clearance to measure GFR within 1 week of the scan session
  Interventions: Other: 3 Tesla multiparametric MR; Other: renal histopathology scoring; Biological: Blood and urine sampling; Biological: Iohexol clearance test
- Acute Kidney Injury: AKI stage 2-3 '3 Tesla multiparametric MR: Renal MRI Scan to assess blood flow, perfusion, oxygenation and microstructure (MR T1 relaxation time and diffusion).
  Each patient will have 3 renal MRI scans. Iohexol clearance test: Blood and urine sampling around scan sessions; this will include routine patient care biochemistry and haematology panel.
  renal histopathology scoring: Blinded fibrosis scoring of renal histopathology (If biopsy performed for clinical indication) urine protein and albumin measurements, stored plasma/serum/urine for subsequent analysis.
  Iohexol clearance to measure GFR within 1 week of the scan session
  Interventions: Other: 3 Tesla multiparametric MR; Other: renal histopathology scoring; Biological: Blood and urine sampling; Biological: Iohexol clearance test

INTERVENTIONS:
Other: 3 Tesla multiparametric MR — Renal MRI Scan to assess blood flow, perfusion, oxygenation and microstructure (MR T1 relaxation time and diffusion). Each patient will have 3 renal MRI scans.
  Other Names: Renal MRI Scan
Other: renal histopathology scoring — Blinded fibrosis scoring of renal histopathology (If biopsy performed for clinical indication)
Biological: Blood and urine sampling — Blood and urine sampling around scan sessions; this will include routine patient care biochemistry and haematology panel,
  urine protein and albumin measurements, stored plasma/serum/urine for subsequent analysis
Biological: Iohexol clearance test — Iohexol clearance to measure GFR within 1 week of the scan session

SUMMARY:
To use Non-invasive MR Imaging of Renal Physiology and structure to assess patients with Acute Kidney Injury (AKI) and Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
Multi centre observational pilot study using novel, contrast free functional renal MRI scans.

A series of functional renal MRI scans will be performed (These scans do not constitute part patients routine clinical care). The results will initially be used to assess renal perfusion and fibrosis in patients with AKI and CKD. Subsequent analysis will be used to identify specific markers on the renal MRI scans that differentiate chronic kidney damage from acute injury to the kidney. Finally results will be used to stratify patients with AKI and CKD into low and high risk of subsequent deterioration in renal function.

AKI Cohort

25 patients with AKI stage 2/3 with or without renal replacement therapy (RRT) will undergo functional renal MRI imaging at day 0, day 90 and day 365.

First Study Scan (Day 0): A functional renal MRI scan will be performed during an admission to hospital with an episode of AKI 2/3. Vital signs and SOFA score will be recorded on the day of the scan.

Renal function assessment will occur± 2 days either side of the scan with an Iohexol clearance test.

Second Study Scan (Day 90): Repeat functional renal MRI imaging will be planned at 90 days (±14 days) after the 1st study scan day.

Renal function assessment will occur±7 days either side of the scan with an Iohexol clearance test.

Third Study Scan (Day 365): The final functional renal MRI imaging will take place 12 months (±30 days) after the 1st study scan day. Renal function assessment will occur±7 days either side of the scan with an Iohexol clearance test.

CKD Cohort:

25 patients with CKD stage 3-4 eGFR 20-59ml/min/1.73m2 will undergo functional renal MRI imaging at day 0, day 7 and day 365.

First Study Scan (Day 0): A functional renal MRI scan will be performed as an outpatient. Vital signs will be recorded on the day of the scan.

Renal function assessment will occur ±7 days either side of the scan with an Iohexol clearance test.

Second Study Scan (Day 7): A functional renal MRI scan will be performed as an outpatient. Vital signs will be recorded on the day of the scan.

Third Study Scan (Day 365): The second functional renal MRI imaging will take place 12 months (±30 days) after the 1st study scan day. Renal function assessment will occur±7 days either side of the scan with an Iohexol clearance test.

ELIGIBILITY:
Inclusion Criteria:

AKI Patients:

* Acute Kidney Injury stage 2/3 (duration >24 hours) including patients requiring renal replacement therapy
* >18 years & < 95 years
* Able to give informed consent

CKD Patients:

* Patients with CKD Stage 3 - 4 (e GFR> 20 and <60 ml/min)
* >18 years & < 95 years
* Able to give informed consent

Exclusion Criteria:

AKI Patients:

* Renal transplant
* Contraindications to MRI e.g. claustrophobia, cardiac pacemaker, metallic fragments or implants
* Pregnancy or breast feeding or intending pregnancy
* Unable to give consent or understand written information
* Pre-existing CKD of any stage as per eGFR
* Obstructive uropathy
* AKI duration <24hrs, in the opinion of the investigator
* Not medically fit for transfer to MRI scan, in the opinion of the clinical team or the investigator
* Iodine allergy
* Patients unable to comply with basic verbal English commands whilst in scanner due to special communication needs

CKD Patients:

* Renal transplant
* Contraindications to MRI e.g. claustrophobia, cardiac pacemaker, metallic fragments or implants
* Pregnancy or breast feeding or intending pregnancy
* Unable to give consent or understand written information
* Unstable CKD; AKI Stage 1 or more or other unplanned hospital admission within the last 90 days
* Iodine allergy
* Patients unable to comply with basic verbal English commands whilst in scanner due to special communication needs

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: secondary care patients
  1. chronic kidney disease stage 3-4 post renal biopsy
  2. Acute kidney injury stage 2-3 during hospital admission
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The difference between volume (mls) MR parameter between healthy volunteers and patients with CKD and AKI | 3 years
  Examining the difference in volume (mls) T1 (ms) between the 3 groups using PRISM, SPSS, Stata and Matlab
The difference between T1 (ms) MR parameter between healthy volunteers and patients with CKD and AKI | 3 years
  Examining the difference in T1 (ms) between the 3 groups using PRISM, SPSS, Stata and Matlab
The difference between Diffusion weighted imaging MR parameter between healthy volunteers and patients with CKD and AKI | 3 years
  Examining the difference in ADC and D(ms) between the 3 groups using PRISM, SPSS, Stata and Matlab

SECONDARY OUTCOMES:
Correlations between structural T1 (ms) and blinded renal biopsy measurements | 3 years
  Sirius red fibrosis scoring (%) Vs T1(ms)
Correlations between structural MR measurement: T1(ms) and creatinine(µmols), | 3 years
  T1 (ms) vs creatinine (µmols)
Correlations between structural diffusion weighted imaging and blinded renal biopsy measurements | 3 years
  Sirius red fibrosis scoring (%) Vs ADC and D (ms)
Correlations between structural MR measurement: diffusion weighted imaging and eGFR mls/min.1.73m | 3 years
  ADC and D (ms) vs eGFR mls/min.1.73m

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, Principal Investigator — univeristy of nottingham; nick selby, Study Chair — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, East Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No